CLINICAL TRIAL: NCT07294781
Title: CircaTime: Effects of Circadian Rhythms on Time Perception During a 36-Hour Constant Routine in Healthy Adults
Brief Title: Circadian Rhythms and Time Perception in Healthy Adults During Constant Wakefulness
Acronym: CircaTime
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Independent Research Fund Denmark (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1-10-72-117-25; 10.46540/4256-00108B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sleep Deprivation; Circadian Rhythm; Healthy Volunteers; Time Perception
Keywords: Circadian rhythms; Constant routine; Extended wakefulness; Sleep loss; Time perception; Subjective time; Psychomotor vigilance task; Dim light melatonin onset; Healthy adults
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: All participants complete a single 36-hour constant-routine protocol with continuous wakefulness under controlled environmental conditions.
Masking Description: Open-label, single-group basic science study; no masking used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Constant Routine Wakefulness (Other): Single-group 36-hour constant-routine protocol with continuous wakefulness. Participants remain in a controlled laboratory environment under low, constant light, with restricted posture and activity, and receive small isocaloric snacks at fixed intervals. Every two hours they complete a standardised test battery assessing time perception, vigilance, mood, and related cognitive and perceptual outcomes.
  Interventions: Behavioral: Constant Routine Wakefulness

INTERVENTIONS:
Behavioral: Constant Routine Wakefulness — Behavioral intervention consisting of approximately 36 hours of continuous wakefulness under constant-routine conditions. Environmental factors (light level, temperature, noise) are held as constant as feasible; posture and activity are standardised; and participants receive small, isocaloric snacks at regular intervals. A repeated cognitive and perceptual test battery is administered every two hours to assess time perception, vigilance, mood, and related functions across the circadian cycle.

SUMMARY:
This study examines how the internal body clock (circadian rhythms) influences the way healthy adults experience time, think, and feel when they stay awake for an extended period. Participants will spend about 36 hours in a controlled sleep laboratory while remaining awake the entire time. Light, posture, food intake, and activity are kept as constant as possible (a "constant routine") so that changes over time mainly reflect the body's internal clock and increasing sleepiness, rather than changes in the environment. Every two hours, participants complete a brief test battery that includes ratings of sleepiness and mood, a reaction-time task, and short tasks that assess how fast or slow time seems to pass, how accurately they can estimate time intervals, how they respond to simple decisions, and how they judge colours. Saliva samples are collected repeatedly to measure melatonin, a hormone that indicates circadian phase. By comparing changes in behaviour, perception, and melatonin levels across the 36-hour wake period, the study aims to identify when during the circadian cycle people are most vulnerable to distortions in time perception and reduced alertness. The findings may help improve scheduling of shift work and other activities that require sustained wakefulness.

DETAILED DESCRIPTION:
Background and Rationale Daily experience of time does not always match clock time: under some conditions time seems to pass faster or slower, and people may misjudge short intervals or deadlines. At the same time, human physiology and cognition are strongly regulated by circadian rhythms, which interact with the build-up of sleep pressure during extended wakefulness. However, it is not well understood how the internal circadian phase and increasing sleepiness jointly shape time perception and related cognitive functions.

The "constant routine" (CR) protocol is a well-established method in circadian research to unmask endogenous rhythmicity. By keeping environmental and behavioural factors as constant as possible while participants remain awake in a semi-recumbent position, the protocol minimises external masking and allows changes over time to be attributed primarily to the underlying circadian system and homeostatic sleep pressure.

Objectives The primary objective is to characterise how time perception (e.g., subjective passage of time and estimation/production of short intervals) varies across the circadian cycle during 36 hours of constant wakefulness. Secondary objectives are to examine how these changes relate to: 1) Biological markers of circadian phase (salivary melatonin), 2) Subjective sleepiness and mood, 3) Objective alertness and vigilance (reaction time), and 4) Simple cognitive decisions and perceptual judgements (e.g., responses to numerical information and colour adjustments).

Study Design This is a single-centre, interventional, basic science study using a within-subject, single-group assignment. Healthy adults attend a screening and briefing visit, followed by one in-laboratory constant-routine session of approximately 36 hours of continuous wakefulness. During the CR, environmental conditions (light, temperature, noise) and posture are controlled, and participants receive small, isocaloric snacks at regular intervals. No drugs, devices, or randomised treatment arms are used; the "intervention" is prolonged wakefulness under constant-routine conditions.

Procedures After eligibility screening and consent, participants complete questionnaires on sleep habits and general health and are instructed to maintain a regular sleep-wake schedule prior to the laboratory visit. For the main CR session, participants arrive at the sleep laboratory in the morning. From that point onward, they remain awake in a controlled setting for about 36 hours. Light is kept at a low, constant level, physical activity is restricted, and posture is standardised as far as feasible.

Every two hours, participants perform a structured test block lasting approximately 45-60 minutes. This block includes: 1) Subjective ratings of sleepiness and mood, 2) A psychomotor vigilance task (reaction-time task), 3) Brief tasks assessing subjective passage of time and the ability to estimate or produce short time intervals, 4) Simple decision-making and estimation tasks, and 5) Perceptual judgements such as colour adjustments.

At regular intervals across the CR, saliva samples are collected to measure melatonin, providing an estimate of individual circadian phase. Vital signs and adverse events are monitored throughout. After the CR, participants are debriefed and provided with recovery sleep arrangements according to local safety procedures.

Outcomes and Analysis Primary outcomes are measures of time perception (e.g., ratings of how fast or slow time seems to pass and accuracy of time interval estimation/production) modelled as a function of circadian phase and hours awake. Secondary outcomes include reaction-time performance, subjective sleepiness and mood ratings, decision-making measures, and colour perception indices. Salivary melatonin profiles are used to determine dim-light melatonin onset (DLMO) and circadian phase position.

Analyses will examine rhythmic changes across the 36-hour protocol and test whether distortions in time perception align with circadian night and with rising sleep pressure. The study is exploratory/basic science in nature and is not designed to evaluate a clinical treatment. Findings are expected to advance understanding of how biological time and psychological time interact, with potential implications for scheduling of shift work, transportation, and other situations requiring sustained wakefulness.

ELIGIBILITY:
Inclusion Criteria:

* Age 23 to 45 years.
* Able and willing to provide written informed consent.
* Fluent in Danish and able to understand study procedures and instructions.
* Generally healthy, as assessed by medical history, screening questionnaires, and basic clinical measures (e.g., blood pressure, heart rate).
* Self-reported regular sleep-wake schedule for at least 4 weeks prior to the laboratory visit (typically 6.5-9 hours of sleep per night, with usual sleep period between approximately 22:00-01:00 and 06:00-09:00).
* Body mass index (BMI) within a non-extreme range (for example, approximately 18.5-30 kg/m²), if required by the study physician.
* No regular night work or rotating shift work during the 3 months before participation.
* No travel across more than 2 time zones in the 2 months before the constant-routine session.
* Willing to abstain from caffeine, nicotine, alcohol, and recreational drugs for the specified washout periods before and during the 36-hour constant-routine session.
* For participants who can become pregnant: negative pregnancy test at screening/arrival and agreement to use reliable contraception for the duration of participation.

Exclusion Criteria:

* Any known or suspected major sleep disorder (e.g., insomnia disorder, obstructive sleep apnoea, restless legs syndrome, narcolepsy), based on self-report or prior diagnosis.
* Current or past major psychiatric or neurological disorders (e.g., major depressive disorder, bipolar disorder, psychotic disorders, epilepsy), unless considered mild and stable and explicitly approved by the study physician.
* Chronic medical conditions that could be worsened by prolonged wakefulness or that might confound outcome measures, such as significant cardiovascular disease, uncontrolled hypertension, diabetes mellitus, severe respiratory disease, or other serious systemic illness.
* Regular use of medications or supplements that may affect sleep, circadian rhythms, melatonin secretion, alertness, or mood (e.g., hypnotics, sedative-hypnotics, melatonin, stimulants, certain antidepressants or beta-blockers), unless a safe washout is possible and approved by the study physician.
* High habitual caffeine intake (for example, >400 mg/day) or nicotine dependence if the participant is unable or unwilling to abstain for the required washout periods.
* Current harmful alcohol use or substance use disorder, or frequent use of recreational drugs.
* Pregnancy or breastfeeding.
* Previous severe adverse reaction to sleep deprivation, extended wakefulness, or similar laboratory protocols.
* Claustrophobia or inability to tolerate prolonged stays in a controlled laboratory environment.
* Any condition or circumstance that, in the judgement of the investigators, would make participation unsafe, interfere with the 36-hour wakefulness protocol, or compromise data quality (e.g., inability to remain awake despite support, strong fear of needles or saliva sampling, or inability to comply with study restrictions).

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Time-Interval Production Error Across 36-Hour Constant Routine | From the beginning of the constant-routine wakefulness session through 36 hours of continuous wakefulness (time-production task completed every 2 hours).
  Mean absolute error (in seconds) between produced and target time intervals on a time-production task. Participants are asked to produce predefined intervals (e.g., several seconds) without external timing cues. For each 2-hour block, time-production error is averaged across trials; analyses model changes in error across circadian phase and hours awake during the 36-hour constant routine.

SECONDARY OUTCOMES:
Subjective Passage-of-Time Ratings Across 36-Hour Constant Routine | From the beginning of the constant-routine wakefulness session through 36 hours of continuous wakefulness (passage-of-time ratings completed every 2 hours).
  Visual analogue scale ratings of how fast or slow time seems to pass "right now" relative to normal (anchors: much slower than normal - much faster than normal). Ratings are collected once per 2-hour test block. For each block, the passage-of-time score is averaged across trials (if multiple ratings) and modelled as a function of circadian phase and hours awake during the 36-hour constant routine.
Psychomotor Vigilance Task (PVT) Median Reaction Time | From the beginning of the constant-routine wakefulness session through 36 hours of continuous wakefulness (PVT completed every 2 hours).
  Median reaction time (milliseconds) on a brief psychomotor vigilance task (PVT) in each 2-hour test block. Participants respond as quickly as possible to visual stimuli presented at random inter-stimulus intervals. For each block, the median reaction time is computed; additional indices such as lapses (responses > 500 ms) may be derived. Changes in PVT performance across the 36-hour constant routine are analysed in relation to circadian phase and hours awake.
Dim Light Melatonin Onset (DLMO) Timing | During the 36-hour constant-routine wakefulness session (salivary melatonin sampled approximately hourly).
  Circadian phase assessed by the timing of dim light melatonin onset (DLMO) derived from repeated salivary melatonin samples collected under constant-routine conditions. DLMO is defined as the clock time at which salivary melatonin concentration first exceeds a predefined threshold (e.g., 3 pg/mL) and remains above that level. This single phase marker per participant is used to align behavioural and perceptual outcomes to individual circadian phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Department of Psychology and Behavioural Sciences, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results will be shared with other researchers upon reasonable request, in accordance with Danish data protection regulations, institutional policies, and ethics approval. Data will be pseudonymised before sharing and no direct identifiers (e.g., name, contact details, personal ID numbers) will be included. Any data elements that could reasonably lead to re-identification in combination with other information will be removed or aggregated where necessary.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified individual participant data and supporting documents will be made available beginning within 12 months after publication of the main results article and will remain available for at least 5 years thereafter.
Access Criteria: De-identified individual participant data (IPD), together with the study protocol, statistical analysis plan, and analytic code, will be available to qualified researchers affiliated with recognised research institutions who submit a methodologically sound proposal and obtain any required ethical or institutional approvals. Requests should describe the planned analyses and data needed. Approved requesters will sign a data use agreement prohibiting re-identification of participants and requiring appropriate data security. Data will be shared via secure transfer or a controlled-access repository approved by Aarhus University.

REFERENCES:
- [Result] Kuriyama K, Uchiyama M, Suzuki H, Tagaya H, Ozaki A, Aritake S, Shibui K, Xin T, Lan L, Kamei Y, Takahashi K. Diurnal fluctuation of time perception under 30-h sustained wakefulness. Neurosci Res. 2005 Oct;53(2):123-8. doi: 10.1016/j.neures.2005.06.006. PMID 16039739
- [Result] Yu C, Van Zuijlen MJP, Spoiala C, Pont SC, Wijntjes MWA, Hurlbert A. Time-of-day perception in paintings. J Vis. 2024 Jan 2;24(1):1. doi: 10.1167/jov.24.1.1. PMID 38165679
- [Result] Hurlbert A, Yu C. Seeing the Light: Perception and Discrimination of Illumination Color. Annu Rev Vis Sci. 2025 Sep;11(1):267-301. doi: 10.1146/annurev-vision-121423-013755. Epub 2025 Aug 5. PMID 40763251
- See also: Sleep & Circadian Psychology Research Unit - Aarhus University (information on research in sleep, circadian rhythms, and time perception) — https://psy.au.dk/en/circadianpsychology